CLINICAL TRIAL: NCT05059444
Title: ORACLE: Observation of ResiduAl Cancer With Liquid Biopsy Evaluation
Acronym: ORACLE
Status: Recruiting | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-MX-003
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bladder Carcinoma; Ureter Carcinoma; Renal Pelvis Carcinoma; Non-small Cell Lung Cancer; Invasive Breast Carcinoma; Cutaneous Melanoma; Esophageal Carcinoma; Gastroesophageal Junction Carcinoma; Gastric Adenocarcinoma; Pancreatic Adenocarcinoma; Squamous Cell Carcinoma of the Head and Neck; Epithelial Ovarian Carcinoma; Fallopian Tube Carcinoma; Endometrial Carcinoma; Renal Cell Carcinoma; Rectal Adenocarcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Endometrial Neoplasms; Carcinoma, Renal Cell; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (12):
- Cohort 1: Muscle invasive carcinoma of the bladder, ureter, or renal pelvis (stage II-III)
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 2: Non-small cell lung cancer (stage IB-III): Cohort 2A: Resectable Cohort 2B: Unresectable
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 3: Invasive breast carcinoma with hormone receptor and HER2 status: Cohort 3A: High-risk HER2+ breast cancer (any ER, PR status allowed); defined as having stage II-III or having residual invasive disease (i.e. non-pathologic complete response) following a neoadjuvant chemotherapy-containing regimen OR Cohort 3B: High-risk triple negative breast cancer (TNBC); defined as having stage II-III or having residual invasive disease (i.e. non-pathologic complete response) following a neoadjuvant chemotherapy-containing regimen OR Cohort 3C: HR-positive/HER2-negative invasive breast carcinoma with either >4 positive axillary lymph nodes or 1-3 positive axillary lymph nodes and at least one of the following: tumor size >5 cm, histologic grade 3, or validated gene expression assay indicating high recurrence risk (OncotypeDx score > 26, MammaPrint high, ProSigna high, EndoPredict high)
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 4: Stage IIB-III cutaneous melanoma or limited (resectable) stage IV melanoma
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 5: Esophageal or gastroesophageal junction carcinoma (stage II-III)
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 6: Gastric adenocarcinoma (stage II-III)
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 7: Pancreatic adenocarcinoma: That is has been surgically resected or is eligible for surgical resection
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 8: Invasive squamous cell carcinoma of the head and neck: Includes stage I-IVB oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, nasal cavity, or paranasal sinus
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 9: High-risk epithelial ovarian or Fallopian tube carcinoma: Defined as FIGO stage IC-III or stage IA-IB that has high grade or clear cell histology.
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 10: High-risk endometrial carcinoma: Defined as FIGO stage II-III.
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 11: High-risk renal cell carcinoma: Defined as high grade (grade 3-4) stage II, stage III or limited (resectable) stage IV treated with curative intent.
  Interventions: Diagnostic Test: Guardant Reveal
- Cohort 12: Pathologically confirmed adenocarcinoma of the rectum: Located up to 15 cm from the anal verge that is undergoing or underwent a preoperative chemotherapy- or immunotherapy-containing regimen

INTERVENTIONS:
Diagnostic Test: Guardant Reveal — Guardant Reveal is a minimal residual disease (MRD) panel for use in recurrence detection of early-stage solid tumors.
  Groups: Cohort 10: High-risk endometrial carcinoma; Cohort 11: High-risk renal cell carcinoma; Cohort 1: Muscle invasive carcinoma of the bladder, ureter, or renal pelvis (stage II-III); Cohort 2: Non-small cell lung cancer (stage IB-III); Cohort 3: Invasive breast carcinoma with hormone receptor and HER2 status; Cohort 4: Stage IIB-III cutaneous melanoma or limited (resectable) stage IV melanoma; Cohort 5: Esophageal or gastroesophageal junction carcinoma (stage II-III); Cohort 6: Gastric adenocarcinoma (stage II-III); Cohort 7: Pancreatic adenocarcinoma; Cohort 8: Invasive squamous cell carcinoma of the head and neck; Cohort 9: High-risk epithelial ovarian or Fallopian tube carcinoma

SUMMARY:
The purpose of ORACLE is to demonstrate the ability of a novel ctDNA assay developed by Guardant Health to detect recurrence in individuals treated for early-stage solid tumors. It is necessary that ctDNA test results are linked to clinical outcomes in order to demonstrate clinical validity for recurrence detection and explore its value in a healthcare environment subject to cost containment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old AND
* Initial treatment is given with curative/radical intent AND
* Are planning to undergo regular follow-up and monitoring for cancer recurrence per standard of care at the enrolling site AND
* Provided written informed consent to participate in the study AND
* Are willing to have de-identified clinical data shared with investigators at regular intervals as outlined in the study protocol and informed consent AND
* Are willing to provide blood samples at enrollment and at subsequent clinical visits coinciding with standard of care follow-up, for up to 5 years as outlined in the study protocol and informed consent AND
* Have at least one Landmark blood sample

Have a histologically confirmed Index Cancer that qualifies for inclusion, defined as:

Primary Study Cohorts

* Cohort 1: Cohort 1: Muscle invasive carcinoma of the bladder, ureter, or renal pelvis (stage II-III),
* Cohort 2: Cohort 2: Non-small cell lung cancer (stage IB-III):

Cohort 2A: Resectable OR Cohort 2B: Unresectable,

* Cohort 3: Invasive breast carcinoma with hormone receptor (e.g. estrogen receptor (ER) and progesterone receptor (PR) expression) and human epidermal growth factor receptor 2 (HER2) status known and one the following:

Cohort 3A: High-risk2 HER2+ breast cancer (any ER, PR status allowed) OR Cohort 3B: High-risk2 triple negative breast cancer (TNBC) OR Cohort 3C: High-risk3 HR-positive/HER2-negative invasive breast carcinoma,

* Cohort 4: Stage IIB-III cutaneous melanoma or limited (resectable) stage IV melanoma treated with curative intent,
* Cohort 5: Esophageal or gastroesophageal junction carcinoma (stage II-III),
* Cohort 6: Gastric adenocarcinoma (stage II-III),
* Cohort 7: Pancreatic adenocarcinoma that is has been surgically resected or is eligible for surgical resection,
* Cohort 8: Invasive squamous cell carcinoma of the head and neck (Includes stage I-IVB oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, nasal cavity, and paranasal sinus cancers),
* Cohort 9: High-risk epithelial ovarian or Fallopian tube carcinoma (Defined as FIGO stage IC-III or stage IA-IB that has high grade or clear cell histology),
* Cohort 10: High-risk endometrial carcinoma (Defined as 2023 FIGO Stage II-III),
* Cohort 11: High-risk renal cell carcinoma (Defined as high grade (grade 3-4) stage II, stage III or limited (resectable) stage IV treated with curative intent)

Exploratory Cohort

* Cohort 12: Pathologically confirmed adenocarcinoma of the rectum (located up to 15 cm from the anal verge) that is undergoing or underwent a preoperative chemotherapy- or immunotherapy- containing regimen

Exclusion Criteria:

* History of allogeneic organ or tissue transplant
* Index cancer has predominantly neuroendocrine histology
* History of another primary cancer diagnosed within 3 years of enrollment, with the exception that in situ cancers, non-melanoma skin carcinomas, localized low- or intermediate risk prostate cancers, and stage I papillary thyroid carcinoma, and participants with bilateral/multifocal tumors within the same organ (for example, bilateral breast cancer) are allowed if diagnosed within 3 years of enrollment
* Known distant metastasis at time of enrollment (with the exception of participants with limited/resectable stage IV cutaneous melanoma or RCC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary study population will include participants with invasive bladder/upper urinary tract carcinoma, NSCLC, breast cancer, cutaneous melanoma, esophageal carcinoma, gastroesophageal junction carcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, squamous cell carcinoma of the head and neck, epithelial ovarian/Fallopian tube carcinoma, endometrial cancer, and renal cell carcinoma (RCC) as per inclusion/exclusion criteria below. Participants with rectal adenocarcinoma undergoing pre-operative systemic chemotherapy/chemoradiotherapy- or immunotherapy-containing regimen are included as an exploratory cohort as per inclusion/exclusion criteria below. Inclusion criteria were selected to enroll participants who are predicted to have >15-20% risk of recurrence within 3 years in order to sufficiently power the study for recurrence events.
Sampling Method: Probability Sample
Enrollment: 2020 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Distant Recurrence Free Interval (D-RFi) | 3 years
  The primary endpoint, distant recurrence-free interval (D-RFi), will be evaluated for each of the primary study cohorts. D-RFi is defined as the time from the end of primary treatment until the time of diagnosis of a distant recurrence of the Index Cancer. Subjects without a distant recurrence will be censored at the time of last follow-up of their Index Cancer.

SECONDARY OUTCOMES:
Sensitivity | 3 years
  Sensitivity defined as the proportion of participants who develop distant recurrence who have ctDNA detected at or before the time of clinical detection of recurrence.
Positive Predictive Value | 3 years
  Positive predictive value (PPV) defined as the proportion of participants who have ctDNA detected at the landmark or any surveillance timepoint who recur (either distally or locally).
Lead Time | 3 years
  Lead time defined as the interval between ctDNA detection and clinical detection of recurrence.

OTHER OUTCOMES:
Recurrence-free interval (RFi) | 3 years
  Recurrence-free interval (RFi) defined as the time from the end of primary treatment until the appearance/occurrence of any recurrence (distant, regional, and/or local) of the Index Cancer. Subjects without recurrence will be censored at the time of last follow-up of their Index Cancer.
Negative predictive value (NPV) | 3 years
  Negative predictive value (NPV) defined as the proportion of participants who have ctDNA not detected who have no evidence of recurrence.
Association with resolution of indeterminate findings | 3 years
  1. The proportion of individuals whose indeterminate finding is ultimately confirmed to be disease recurrence who have ctDNA detected at the initial time the indeterminate finding is identified and
  2. The proportion of ctDNA not detected participants whose indeterminate findings is ultimately confirmed to be benign.
Sensitivity for local recurrence | 3 years
  Sensitivity for local recurrence defined as the proportion of participants who have localized recurrence (e.g., in the absence of distant metastasis) who have ctDNA detected at or before the time of clinical detection of a localized recurrence; using landmark and serial timepoints.
Index Cancer-Specific Survival (ICSS) | 3 years
  Index Cancer-Specific Survival (ICSS) defined as the time from the date of diagnosis until the date of death from the subject's Index Cancer. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Overall Survival (OS) | 3 years
  Overall Survival (OS) defined as the time from the date of diagnosis until the date of death from any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Rate of ctDNA clearance with adjuvant chemotherapy | 3 years
  Rate of ctDNA clearance with adjuvant chemotherapy defined as the proportion of patients who have ctDNA detected at the pre-enrollment timepoint whose ctDNA becomes undetectable at the Landmark timepoint.
Association of ctDNA detection status with pathologic response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Guardant Health, Inc.
Locations (57):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - University of California, San Diego, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Redwood City, Redwood City, California
  - Sutter Institute for Medical Research, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Memorial Healthcare System, Hollywood, Florida
  - The Oncology Institute of Hope & Innovation, Lakeland, Florida
  - Tulane Cancer Center, New Orleans, Louisiana
  - Christus Highland/ Boniol, Shreveport, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mayo Clinic (Rochester), Rochester, Minnesota
  - Astera Cancer Care, East Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC- Chapel Hill, Chapel Hill, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Crozer-Keystone Health System, Broomall, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - DHR Health Advance Care Center, Edinburg, Texas
  - The Center for Cancer and Blood Disorders, Forth Worth, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
- France (5):
  - CHU Besançon, Besançon
  - Hôpital Franco-Britannique, Levallois-Perret
  - Institut Paoli-Calmettes, Marseille
  - Ambroise Paré-Hartmann, Neuilly
  - APHP Tenon Hospital - Sorbonne, Paris
- Germany (3):
  - Asklepios Klinik Altona, Hamburg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Ludwig Maximilian University Munich, Munich
- Italy (3):
  - Instituto Romagnolo per lo Studio dei Tumori "Dino Amadori" IRCCS IRST, SrL, Meldola
  - Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Agostino Gemelli, Roma
- Spain (13):
  - Hospital Teresa Herrera (C.H.U.A.C), A Coruña
  - Vall Hebron Institute of Oncology, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - ICO Institut Catala d'Oncologia, Barcelona
  - Instituto Catalan de Oncologia de Girona, Girona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - CIOSS HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - CCS Hospital Universitari Parc Taulí, Sabadell
  - Hospital Clinico de Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No